CLINICAL TRIAL: NCT04534855
Title: A Phase II Single Arm Clinical Study of Treprilimab in the Treatment of Local Recurrent/Residual Nasopharyngeal Carcinoma After Re-irradiation
Brief Title: A Phase II Clinical Study of Treprilimab in the Treatment of Recurrent Nasopharyngeal Carcinoma After Re-irradiation
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Fei Han, Deputy Director of radiotherapy Department, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: B2020-154-01
Record Dates: First submitted 2020-08-25; First posted 2020-09-01 (Actual); Last update posted 2020-09-01 (Actual); Status verified 2020-08

CONDITIONS: Nasopharyngeal Carcinoma
Keywords: Treprilimab,recurrent/residual NPC
MeSH Terms: conditions — Nasopharyngeal Carcinoma

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treprilimab treatment group (Experimental): Treprilimab 240mg ivdrip Q3W until progression or unacceptable toxicity
  Interventions: Drug: Treprilimab

INTERVENTIONS:
Drug: Treprilimab — Treprilimab 240mg Q3W until progression or unacceptable toxicity

SUMMARY:
To establish the antitumor activity and safety of the anti-programmed death 1 receptor monoclonal antibody, Treprilimab, in patients with local recurrent/residual nasopharyngeal carcinoma after re-irradiation.Patients with local recurrent/residual NPC after re-irradiation were treated with Treprilimab until disease progression or unacceptable toxicity. The primary end point was objective response rate (ORR) and secondary end points included survival and toxicity.The sample size of this study was estimated on the assumption that response rates (RRs) to Treprilimab should be around 25%,based on a report that was available at the time this study was planned.Furthermore, the RR to noncytotoxic, experimental agents such as pazopanib and cetuximab in similarly pretreated patient cohorts was approximately 5% to 10%. This study's design was based on the modiﬁed Simon two-stage optimal design (α=0.05，β=0.2,n1=2/22,n2=7/40). If two responses were observed during the ﬁrst stage, enrollment was continued until a total of 40 patients was reached.

DETAILED DESCRIPTION:
To establish the antitumor activity and safety of the anti-programmed death 1 receptor monoclonal antibody, Treprilimab, in patients with local recurrent/residual nasopharyngeal carcinoma after re-irradiation.Patients with local recurrent/residual NPC after re-irradiation were treated with Treprilimab until disease progression or unacceptable toxicity. The primary end point was objective response rate (ORR) and secondary end points included survival and toxicity.The sample size of this study was estimated on the assumption that response rates (RRs) to Treprilimab should be around 25%,based on a report that was available at the time this study was planned.Furthermore, the RR to noncytotoxic, experimental agents such as pazopanib and cetuximab in similarly pretreated patient cohorts was approximately 5% to 10%. This study's design was based on the modiﬁed Simon two-stage optimal design (α=0.05，β=0.2,n1=2/22,n2=7/40). If two responses were observed during the ﬁrst stage, enrollment was continued until a total of 40 patients was reached. The target lesions had to be measurable by the Response Evaluation Criteria in Solid Tumors (RECIST). Radiologic assessments were performed every 8 weeks for 6 months and then every 12 weeks thereafter. Eligible patients were treated with Treprilimab at a dosage of 240mg intravenously every 3 weeks until they experienced disease progression or unacceptable toxicity. The primary end point of this study was objective response by the RECIST criteria , and the secondary end points were overall survival (OS), progression-free survival (PFS), duration of response and toxicity.

ELIGIBILITY:
Inclusion Criteria:

* ages from 18 years to 65 years.
* Histologically confirmed local recurrent/residual Nasopharyngeal carcinoma with previous re-irradiation.
* measurable disease at baseline on the basis of RECIST v1.1.
* Eastern Cooperative Oncology Group performance status of 0 or 1.
* adequate organ function.
* anticipate survival≥3 months.

Exclusion Criteria:

* a diagnosis of immuno deﬁciency or systemic corticosteroid therapy within 14 days of study start.
* prior anticancer monoclonal antibody therapy within 4 weeks of study start.
* any anticancer therapy within 4 weeks preceding the study start.
* therapy with any other immune checkpoint inhibitor.
* active autoimmune disease, interstitial lung disease, known additional malignancy that was progressing or that required active treatment.
* not received platinum based chemotherapy previously.
* confirmed systemic metastasis
* HBV positive and Child-Pugh B or C cirrhosis
* HCV positive and Child-Pugh B or C cirrhosis

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2020-09-01 (Estimated); Primary Completion 2022-09-01 (Estimated); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
objective response rate | Response was assessed by magnetic resonance imaging every 8 weeks for the ﬁrst 6 months and every 12 weeks thereafter.
  the proportion of patients with conﬁrmed complete response or partial response (PR) per RECIST v1.1

SECONDARY OUTCOMES:
PFS | time from enrollment to the ﬁrst documented progression of disease or death from any cause)
  progression free survival
OS | time from enrollment to death from any cause
  overall survival
Number of participants with treatment-related adverse events | through the study and for 30 days after treatment discontinuation (90 days for serious AEs).
  Number of participants with treatment-related adverse events as assessed by CTCAE v4.0

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code

REFERENCES:
- [Background] Ma BBY, Lim WT, Goh BC, Hui EP, Lo KW, Pettinger A, Foster NR, Riess JW, Agulnik M, Chang AYC, Chopra A, Kish JA, Chung CH, Adkins DR, Cullen KJ, Gitlitz BJ, Lim DW, To KF, Chan KCA, Lo YMD, King AD, Erlichman C, Yin J, Costello BA, Chan ATC. Antitumor Activity of Nivolumab in Recurrent and Metastatic Nasopharyngeal Carcinoma: An International, Multicenter Study of the Mayo Clinic Phase 2 Consortium (NCI-9742). J Clin Oncol. 2018 May 10;36(14):1412-1418. doi: 10.1200/JCO.2017.77.0388. Epub 2018 Mar 27. PMID 29584545
- [Background] Hsu C, Lee SH, Ejadi S, Even C, Cohen RB, Le Tourneau C, Mehnert JM, Algazi A, van Brummelen EMJ, Saraf S, Thanigaimani P, Cheng JD, Hansen AR. Safety and Antitumor Activity of Pembrolizumab in Patients With Programmed Death-Ligand 1-Positive Nasopharyngeal Carcinoma: Results of the KEYNOTE-028 Study. J Clin Oncol. 2017 Dec 20;35(36):4050-4056. doi: 10.1200/JCO.2017.73.3675. Epub 2017 Aug 24. PMID 28837405
- [Background] Chan AT, Hsu MM, Goh BC, Hui EP, Liu TW, Millward MJ, Hong RL, Whang-Peng J, Ma BB, To KF, Mueser M, Amellal N, Lin X, Chang AY. Multicenter, phase II study of cetuximab in combination with carboplatin in patients with recurrent or metastatic nasopharyngeal carcinoma. J Clin Oncol. 2005 May 20;23(15):3568-76. doi: 10.1200/JCO.2005.02.147. Epub 2005 Apr 4. PMID 15809453
- [Background] Zhou Y, Miao J, Wu H, Tang H, Kuang J, Zhou X, Peng Y, Hu D, Shi D, Deng W, Cao X, Zhao C, Xie C. PD-1 and PD-L1 expression in 132 recurrent nasopharyngeal carcinoma: the correlation with anemia and outcomes. Oncotarget. 2017 Apr 19;8(31):51210-51223. doi: 10.18632/oncotarget.17214. eCollection 2017 Aug 1. PMID 28881642